CLINICAL TRIAL: NCT01677585
Title: PROMUS Element™ China Post-Approval Study
Brief Title: Post-Approval Study of PROMUS Element™ in China
Acronym: PEChina
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2288
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compile real-world clinical outcomes data for the PROMUS Element™ and PROMUS Element™ Plus Everolimus-Eluting Coronary Stent System (PROMUS Element and PROMUS Element Plus Stent System) in routine clinical practice in China.

DETAILED DESCRIPTION:
Everolimus-eluting stents have been studied extensively in ongoing clinical studies. The safety and effectiveness of the everolimus drug and polymer combination have been studied extensively in the SPIRIT Clinical Trial Program. The PROMUS Element stent is currently being studied in the PLATINUM Clinical Trial Program. The PROMUS Element stent is also being evaluated in PROMUS Element Plus US post-approval studies and the ongoing Platinum China study. This study is designed to provide post-market surveillance information on the PROMUS Element™ and PROMUS Element™ Everolimus-Eluting Coronary Stent System (PROMUS Element and PROMUS Element Plus Stent System) after it has been approved by SFDA (State of Food and Drug Administration) in China. The study will evaluate clinical outcomes for subjects receiving the PROMUS Element and PROMUS Element plus stents over 5 years in a real world setting according to post approval requirements from SFDA.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject understands and provides written informed consent
* Subject who is clinically indicated and will have an attempt of at least one PROMUS Element stent OR Subject who is clinically indicated and was implanted with at least one PROMUS Element stent
* Subject is willing to comply with all protocol-required follow-up evaluation

Exclusion Criteria:

* Exclusion criteria is not required in the PROMUS Element China Post-Approval study which is an "all comers" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are candidates for coronary artery stenting, signed the informed consent form and eligible to receive a PROMUS Element stent will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate | 12-month
  The primary endpoint is the 12-month target lesion failure (TLF) rate, defined as any ischemia-driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Professor, Principal Investigator — Second Affliated Hosptial Zhejiang University College of Medicine
Locations (1):
- Second Affliated Hosptial Zhejiang University College of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No